CLINICAL TRIAL: NCT04269044
Title: The Efficacy of a Novel, Non-contact EKG in the NICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Andrew Gostine, MD, Anesthesiologist and Intensivist, Northwestern Medicine
Other Study IDs: 20-006-LFH
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Electrocardiogram Electrode Site Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: non-contact EKG — ultra-sensitive, non-contact EKG pad will be placed beneath the infant
  Other Names: standard, contact EKG

SUMMARY:
We will be comparing a novel, non-contact EKG waveform and heart rate to the standard of care, contact-based EKG waveform and heart rate in neonates, who have sensitive skin.

ELIGIBILITY:
Inclusion Criteria:

* Apgar at 5 min >/= 7
* Admitted to the NICU
* Indication for standard EKG monitoring

Exclusion Criteria:

* Apgar < 7 at 5 min
* Not in the NICU
* Not being monitored with standard EKG monitors

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will be studying neonates in the NICU. They have sensitive skin and thus a suspected benefit from switching to a non-contact EKG
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
difference in heart rate | 1 hour
  we will compare the two heart rate figures from both EKG sources

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Lake Forest Hospital, Lake Forest, Illinois, United States

IPD SHARING:
Plan to Share IPD: No